CLINICAL TRIAL: NCT03537326
Title: Study to Detect Oral Administration of Budesonide in Women.
Acronym: WADA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Julian Mateus, Clinical Pharmacologist (Md), Parc de Salut Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IMIMFTCL/DACORSIN/3; 2017-004839-37 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: doping
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Healthy women, aged between 18 and 45 years old, weighing between 50 and 75 kg and with BMI included between 19 and 27 kg/m².
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Budesonide (Experimental): Healthy women, aged between 18 and 45 years old, with weigh between 50 and 75 kg and with IMC included between 19 and 27 kg/m². Patients will be given, on an empty stomach since 10 hours minimum, a single dose of 3 mg of Budesonide, in the form of Entocord ® tablets. After that, they will remain under medical control for at least an hour, and then will be back home with instructions to collect urine samples at defined times, during 4 days.
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Patients will be given, on an empty stomach since a minimum of 10 hours, a single dose of 3 mg of Budesonide, in the form of Entocord® capsuls. After that, they will remain under medical control for at least an hour, and then will be back home with instructions to collect urine samples at defined times, during 4 days.
  Other Names: Entocord® modified release capsule, 3 mg single-dose

SUMMARY:
This study aims at identifying analysis strategies to detect oral administration of Budesonide in women; in order for them to be used by the accredited laboratories of the Worl Anti-Doping Agency (WADA).

DETAILED DESCRIPTION:
This clinical trial aims at studying the budesonide metabolism of women. The objective is to identify analysis strategies to detect oral administration of Budesonide in women. In order to use them in the accredited laboratories of the Worl Anti-Doping Agency (WADA).

This study will also help with defining the referential levels of this way of administration. Also, it will be used to test the safety and tolerability of the medication used.

For this, will be collected at precise times after the oral administration of the medication, the concentrations in urines of the metabolite o budesonide : the 6bêta-hydroxy-budesonide, of budesonide itself, of other metabolites. These concentrations will be compare to the ones in the basal samples of subject's urines.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers aged from 18 to 45 years.
* Understand and accepting the procedures of the trial and sign an informed consent.
* Have a history and physical exams that show that there is no organic or psychiatric problems.
* The ECG, and the general blood and urine analyses done before the trial, have to be in the normal limits. Punctual or minor variations outside limits could be accepted if, according to the Main Investigator and regarding the state of science, they don't have clinical impact, can't present a risk for the subjects and don't interfere in the medication evaluation. These variations and their non-relevance will be specifically justified in writing.
* The subjects must weigh between 50 and 75kg, with a BMI between 19 and 27 kg/m2.

Exclusion Criteria:

* Don't fulfilling one or several inclusion criteria.
* Have a medical history of allergy, idiosyncrasy, hypersensibility or adverse reactions to corticoids or the medication excipients. Have a medical history of serious adverse reaction to some medication.
* Subjects with contraindication to treatments with the trial's medication (according to the respective data sheet).
* Medical history or clinical evidence of gastrointestinal, hepatic or renal issue; or other types of issue that could suppose a deterioration of medication abortion, distribution, metabolism or excretion, or that could suggest gastrointestinal irritation by any medication.
* Medical history or clinical evidence of issue that would be psychiatric, alcoholism, medication or drugs abuse, or usual consumption of psychoactive medication.
* Participate in a clinical trial involving medication in the last 3 months before the beginning of the trial.
* Have done a blood donation during the last 3 months preceding of the study, if it's necessary to draw blood for the study.
* Have suffered from an organic illness or major emergency during the 6 months preceding the trial.
* Medical history or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, haematologic or neurologic disease; or other acute or chronic illness that, according to the Main Investigator or collaborators designated by him, could present a risk for the subjects or interfere in the study objectives. Especially osteoporosis, high blood pressure, Cushing syndrome, diabetes mellitus and viral infections such as herpes or varicella.
* Having regularly taken medication during the month preceding the study, excepted vitamins, herbal medication or dietetics complementation that, according to the Main Investigator or collaborators designated by him, could present a risk for the subjects or interfere in the study objectives. The intake of a single-dose symptoms medication during the previous week will not be an exclusion criterion if it is considered as completely eliminated the day beginning the experimental session.
* Smoke more than 20 cigarets per day during the last 3 months before the study.
* Consume more than 20g of alcohol per day.
* Consume more than 5 cafés, teas, cola drinks or other stimulating drinks or with xanthine per day in the 3 months preceding the start of the study.
* Not being able to understand the nature of the study and procedures that it implies to follow.
* Have a positive serology for B or C hepatitis or HIV.
* Being pregnant or breastfeeding and don't use reliable means of contraception during the study.
* Take hormonal contraceptives (oral, topic, injectable or vaginal).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
6β-hydroxy-budesonide urine concentration. | 0-4 hr (hours) ; 4-8 hr ; 8-12 hr ; 12-24 hr ; 24-36 hr ; 36-48 hr ; 48-72 h ; 72-96 hr after administration
  Many defined times after the oral administration of Entocord®, urine sample will be collected by the subjects and then analysed in laboratory to determine 6β-hydroxy-budesonide concentration.

SECONDARY OUTCOMES:
Medication and other metabolites urine concentrations. | 0-4 hr ; 4-8 hr ; 8-12 hr ; 12-24 hr ; 24-36 hr ; 36-48 hr ; 48-72 hr ; 72-96 hr after administration
  Many defined times after the oral administration of Entocord®, urine samples will be collected by the subjects and then analysed in laboratory to determine concentrations of Entocord® and other metabolites of budesonide.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Ventura Alemany, Pharmacéutic, Principal Investigator — Laboratorio Antidopaje de Catalunya.
Locations (1):
- IMIM, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai TR. Glucocorticosteroid treatment of asthma. Can Fam Physician. 1995 Nov;41:1921-7. PMID 8563509
- [Background] Czock D, Keller F, Rasche FM, Haussler U. Pharmacokinetics and pharmacodynamics of systemically administered glucocorticoids. Clin Pharmacokinet. 2005;44(1):61-98. doi: 10.2165/00003088-200544010-00003. PMID 15634032
- [Background] Deventer K, Delbeke FT. Validation of a screening method for corticosteroids in doping analysis by liquid chromatography/tandem mass spectrometry. Rapid Commun Mass Spectrom. 2003;17(18):2107-14. doi: 10.1002/rcm.1157. PMID 12955741
- [Background] Duclos M. [Use and abuse of anabolic steroids and glucocorticoids in sport]. Ann Endocrinol (Paris). 2007 Sep;68(4):308-14. doi: 10.1016/j.ando.2007.06.022. Epub 2007 Aug 8. No abstract available. French. PMID 17689473
- [Background] Fluri K, Rivier L, Dienes-Nagy A, You C, Maitre A, Schweizer C, Saugy M, Mangin P. Method for confirmation of synthetic corticosteroids in doping urine samples by liquid chromatography-electrospray ionisation mass spectrometry. J Chromatogr A. 2001 Aug 10;926(1):87-95. doi: 10.1016/s0021-9673(01)01065-2. PMID 11554422
- [Background] Ho EN, Leung DK, Wan TS, Yu NH. Comprehensive screening of anabolic steroids, corticosteroids, and acidic drugs in horse urine by solid-phase extraction and liquid chromatography-mass spectrometry. J Chromatogr A. 2006 Jul 7;1120(1-2):38-53. doi: 10.1016/j.chroma.2006.03.089. Epub 2006 May 2. PMID 16631183
- [Background] Matabosch X, Pozo OJ, Perez-Mana C, Farre M, Marcos J, Segura J, Ventura R. Discrimination of prohibited oral use from authorized inhaled treatment of budesonide in sports. Ther Drug Monit. 2013 Feb;35(1):118-28. doi: 10.1097/FTD.0b013e3182787b20. PMID 23318282
- [Background] Matabosch X, Pozo OJ, Perez-Mana C, Farre M, Marcos J, Segura J, Ventura R. Identification of budesonide metabolites in human urine after oral administration. Anal Bioanal Chem. 2012 Aug;404(2):325-40. doi: 10.1007/s00216-012-6037-0. Epub 2012 May 10. PMID 22573060
- [Background] Spyridaki MH, Kiousi P, Vonaparti A, Valavani P, Zonaras V, Zahariou M, Sianos E, Tsoupras G, Georgakopoulos C. Doping control analysis in human urine by liquid chromatography-electrospray ionization ion trap mass spectrometry for the Olympic Games Athens 2004: determination of corticosteroids and quantification of ephedrines, salbutamol and morphine. Anal Chim Acta. 2006 Jul 28;573-574:242-9. doi: 10.1016/j.aca.2006.04.042. Epub 2006 Apr 27. PMID 17723530
- [Background] Touber ME, van Engelen MC, Georgakopoulus C, van Rhijn JA, Nielen MW. Multi-detection of corticosteroids in sports doping and veterinary control using high-resolution liquid chromatography/time-of-flight mass spectrometry. Anal Chim Acta. 2007 Mar 14;586(1-2):137-46. doi: 10.1016/j.aca.2006.09.058. Epub 2006 Oct 5. PMID 17386705
- [Result] Andersen JH, Hansen LG, Pedersen M. Optimization of solid phase extraction clean up and validation of quantitative determination of corticosteroids in urine by liquid chromatography-tandem mass spectrometry. Anal Chim Acta. 2008 Jun 9;617(1-2):216-24. doi: 10.1016/j.aca.2008.02.070. Epub 2008 Mar 27. PMID 18486661